CLINICAL TRIAL: NCT00189280
Title: Open Study to Evaluate the Efficacy and Tolerance of Imiquimod 5% Cream for the Treatment of a Large and/or Multiple Superficial Basal Cell Carcinoma.
Brief Title: Aldara for the Treatment of Large and/or Multiple sBCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Elena Rizova, MD, Medical and Scientific Affairs, Europe & MENA, Laboratoires 3M Santé
Organization: Viatris Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1475-IMIQ
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2022-02-22 (Actual); Status verified 2008-09

CONDITIONS: Carcinoma, Basal Cell
Keywords: Aldara, sBCC
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Imiquimod

ARMS (1):
- imiqimod 5% cream (Experimental)
  Interventions: Drug: Imiquimod

INTERVENTIONS:
Drug: Imiquimod — cream 5%, 5 days out of seven, for 6 weeks

SUMMARY:
BCC is the most common form of skin cancer. Current treatment is often surgery but this can be limited by the number of lesions, their location the age of the patient or the potential cosmetic outcome. The purpose of this study is to evaluate the effectiveness of imiquimod, on a non surgical treatment, in subjects with multiple of large sBCCs.

ELIGIBILITY:
Inclusion Criteria:

* One or more sBCC on torso, neck or face
* Total surface area <= 40 sq cm

Exclusion Criteria:

* Pregnancy or women who are breastfeeding
* Xeroderma pigmentosum, albinism, epidermodysplasia verruciformis, any genetic anomaly accompanied by skin tumors
* Metatypical, adnexal, or sclerodermiform carcinomas
* Current or other previous malignant skin tumor (epidermoid carcinoma, melanoma) in the region of the current lesion
* Known HIV positive serology
* Skin tumor that is already or highly likely to become metastatic
* Presence of a clinically significant anomaly or illness (immunological, cardiovascular, pulmonary, hematological, neurological, hepatic, renal, endocrine, gastrointestinal, collagenous)
* Previous organ transplant history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2003-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Clinical clearance of sBCC | 12 or 16 weeks after treatment

SECONDARY OUTCOMES:
Reduction in size of tumour | 12 or 16 weeks after treatment
Rate of clearance, Cosmetic outcome | 12 or 16 weeks after treatment
Sustained clearance rate over 3 year follow-up | 3 years after treatment
Tolerability & QoL | 12 or 16 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Professeur Bedane, Principal Investigator — Service de DermatologieHôpital Dupuytren, LIMOGES
Locations (1):
- Service de DermatologieHôpital Dupuytren, Limoges, France